CLINICAL TRIAL: NCT00668642
Title: Effect of Dutasteride on Androgen-Response Gene Expression During the Tumor Regrowth Phase of Intermittent Androgen Ablation Therapy in Patients With Advanced Prostate Cancer
Brief Title: Effect of Dutasteride on Androgen-Response Gene Expression in Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: University of Chicago (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Daniel Shevrin, Principal Investigator, Division of Hematology/Oncology, Endeavor Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EH07-109
Record Dates: First submitted 2008-04-28; First posted 2008-04-29 (Estimated); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Dutasteride During First Off-Cycle (Experimental): Arm A patients received dutasteride (0.5 mg/day) during the first off-cycle and received placebo during the second off-cycle
  Interventions: Drug: Dutasteride
- B: Placebo During First Off-Cycle (Placebo Comparator): Arm B patients received placebo during the first off-cycle and received dutasteride (0.5 mg/day) during the second off-cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride — 0.5 mg capsule given orally on daily basis
  Other Names: Avodart
  Arms: A: Dutasteride During First Off-Cycle
Drug: Placebo — Identical placebo
  Arms: B: Placebo During First Off-Cycle

SUMMARY:
The purpose of this study is to determine if the drug dutasteride increases expression of genes that slow the growth of prostate cancer during treatment with intermittent androgen ablation therapy (hormone therapy).

DETAILED DESCRIPTION:
We have shown in a murine model of treatment with intermittent androgen ablation therapy of prostate cancer that when dutasteride is given during the regrowth phase (off-phase) of intermittent therapy, that tumor growth is inhibited and that survival is improved. We have also shown that testosterone is a more potent inducer of certain tumor suppressor androgen response genes than dihydrotestosterone. In this murine model, we showed that use of a 5-alpha reductase inhibitor (dutasteride) resulted in significant hyperinduction of the U19 tumor suppressor androgen response gene during the regrowth phase of treatment. In the current clinical trial, we will determine if use of dutasteride in men with advanced prostate cancer during the off-phase of intermittent androgen ablation therapy will also result in hyperinduction of these tumor suppressor androgen response genes. Gene expression will be measured in tumor tissue obtained by prostate biopsies during the off-phase when the testosterone level has normalized. Prostate-specific antigen (PSA) levels will also be measured to determine the PSA doubling time during the off-phase to determine the effect of dutasteride on PSA kinetics.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer
* Patients are hormone-naive
* Patients either to begin androgen ablation therapy with luteinizing hormone-releasing hormone (LHRH) agonist or already receiving therapy with LHRH agonist
* Advanced prostate cancer with either positive pelvic nodes or bone/visceral metastasis
* Must have an intact prostate (no previous surgery or XRT)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Recovery from any major infection or surgical procedure
* Signed informed consent

Exclusion Criteria:

* Known intolerance or allergy to dutasteride
* Concomitant chemotherapy, biologic therapy, or XRT to prostate
* Bilateral orchiectomy
* Prior malignancy within 5 years of registration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Shevrin, MD, Principal Investigator — Endeavor Health
Locations (3):
- United States (3):
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago Hospitals and Clinics, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 participants enrolled and all received initial treatment with anti-androgen therapy (AAT) for planned 8 months (on-cycle 1). 7 participants progressed during this treatment, so 13 participants proceeded with randomization.
Period: First Off-cycle
Arm/Group | A: Dutasteride During First Off-Cycle | B: Placebo During First Off-Cycle
Started | 7 | 6
Research Biopsy (A research biopsy of the prostate was planned at end of off-cycle 1 to determine expression of U19 tumor suppressor gene) | 4 | 3
Completed | 6 | 6
Not Completed | 1 | 0
Not completed — Cancer progression | 1 | 0
Period: Second AAT Treatment (On-cycle 2)
Arm/Group | A: Dutasteride During First Off-Cycle | B: Placebo During First Off-Cycle
Started | 6 | 6
Completed | 4 | 5
Not Completed | 2 | 1
Not completed — Cancer progression | 2 | 1
Period: Second Off Treatment (Off-cycle 2)
Arm/Group | A: Dutasteride During First Off-Cycle | B: Placebo During First Off-Cycle
Started | 4 | 5
Research Biopsy (A research biopsy of the prostate was planned at end of off-cycle 2 to determine expression of U19 tumor suppressor gene) | 2 | 2
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 20 participants enrolled to study and received initial AAT treatment for 8 months (on-cycle 1)
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Dutasteride During First Off-Cycle | B: Placebo During First Off-Cycle | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 67 (20) | 67 (20) | 67 (20)
Sex: Female, Male [Count of Participants; unit: Participants] — Male participants only
  Participants
    Female | 0 | 0 | 0
    Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relative Expression of U19 Gene in Tumor From Prostate Gland During First Off-cycle.
Description: Calculation of the level of gene expression of the U19 tumor suppressor gene compared between the 2 arms at the end of "off-treatment" cycle 1.
Time Frame: At the end of off-cycle 1 defined by when the testosterone level reaches normal (approximately 6 months)
Population: Only patients from each arm with biopsies at the end of off-cycle 1 are included.
Measure: Mean (Standard Deviation); unit: Relative expression
Arm/Group | A: Dutasteride During First Off-Cycle | B: Placebo During First Off-Cycle
Number analyzed (Participants) | 4 | 3
Relative expression | 0.24 (0.5) | 0.28 (0.45)

2. Secondary Outcome: Determination of Prostate-specific Antigen (PSA) Doubling Time During First Off-cycle
Description: Calculation of number of months when baseline PSA doubles compared between the 2 arms at the end of "off-treatment" cycle 1.
Time Frame: At month 9 and ongoing monthly until end of off-cycle 1 defined by when the testosterone level reaches normal (approximately 6 months)
Population: Only patients from each arm with biopsies at the end of off-cycle 1 are included.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | A: Dutasteride During First Off-Cycle | B: Placebo During First Off-Cycle
Number analyzed (Participants) | 4 | 3
Months | 1.42 (0.8) | 1.56 (0.9)

ADVERSE EVENTS:
Arm/Group | A: Dutasteride During First Off-Cycle | B: Placebo During First Off-Cycle
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Dutasteride During First Off-Cycle (N=7) | B: Placebo During First Off-Cycle (N=6)
Decrease in libido (Reproductive system and breast disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No